CLINICAL TRIAL: NCT03613818
Title: Efficacy of a Web-Based Alcohol Intervention for High School Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boise State University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Diana Doumas, Distinguished Professor, Boise State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 023880; R21AA023880 (NIH)
Record Dates: First submitted 2018-07-30; First posted 2018-08-03 (Actual); Results first posted 2021-04-01 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Underage Drinking
MeSH Terms: conditions — Underage Drinking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- eCHECKUP TO GO (Experimental): Brief, web-based alcohol intervention
  Interventions: Behavioral: eCHECKUP TO GO
- Control (No Intervention): Assessment only

INTERVENTIONS:
Behavioral: eCHECKUP TO GO — eCHECKUP TO GO is a personalized normative feedback intervention intended to help participants make better choices about alcohol use by changing beliefs about alcohol, alcohol expectancies, and perceptions of peer drinking
  Arms: eCHECKUP TO GO

SUMMARY:
This study evaluates the efficacy of the eCHECKUP TO GO as an intervention to reduce underage drinking and the associated negative consequences among high school seniors. The aim of this project is to provide a brief, low cost intervention that can be easily disseminated as a school-based intervention to address this important public health problem.

ELIGIBILITY:
Inclusion Criteria:

* Senior enrolled in high school sites

Exclusion Criteria:

* none

Ages: 16 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 311 (Actual)
Dates: Start 2018-09-15 (Actual); Primary Completion 2019-04-01 (Actual); Study Completion 2019-04-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Diana Doumas, PhD, Principal Investigator — Boise State Univeristy
Locations (1):
- Boise State University, Boise, Idaho, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Doumas DM, Esp S, Turrisi R, Bond L, Flay B. Efficacy of the eCHECKUP TO GO for High School Seniors: Sex Differences in Risk Factors, Protective Behavioral Strategies, and Alcohol Use. J Stud Alcohol Drugs. 2020 Mar;81(2):135-143. doi: 10.15288/jsad.2020.81.135. PMID 32359042
- [Derived] Doumas DM, Esp S, Turrisi R, Bond L, Glenn SD. A randomized controlled trial testing the efficacy of the eCHECKUP TO GO on drinking games participation and behavior among high school seniors. Addict Behav. 2025 Jan;160:108183. doi: 10.1016/j.addbeh.2024.108183. Epub 2024 Sep 30. PMID 39388851
- [Derived] Doumas DM, Esp S, Turrisi R, Bond L. A Randomized Controlled Trial of the eCHECKUP to GO for High School Seniors across the Academic Year. Subst Use Misuse. 2021;56(13):1923-1932. doi: 10.1080/10826084.2021.1958862. Epub 2021 Aug 4. PMID 34347564

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | eCHECKUP TO GO | Control
Started | 174 | 137
Completed | 137 | 110
Not Completed | 37 | 27

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | eCHECKUP TO GO | Control | Total
Number analyzed (Participants) | 174 | 137 | 311
Age, Continuous [Mean (Standard Deviation); unit: years] | 17.13 (0.46) | 17.13 (0.45) | 17.13 (0.45)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 100 | 73 | 173
  Male | 74 | 64 | 138
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 152 | 112 | 264
  Hispanic/Latino | 6 | 9 | 15
  Asian | 7 | 7 | 14
  Black/African-American | 1 | 4 | 5
  American Indian/Alaska Native | 2 | 2 | 4
  Native Hawaiian/Pacific Islander | 2 | 0 | 2
  Other | 4 | 3 | 7
Region of Enrollment [Number; unit: participants]
  United States | 174 | 137 | 311

OUTCOME MEASURES:

1. Primary Outcome: Weekly Drinking
Description: Daily Drinking Questionnaire
  Weekly drinking was assessed with the question "Given that it is a typical week, please write the number of drinks you probably would have each day." A response scale is provided for each day of the week (e.g., Monday__, Tuesday__, etc.)." Weekly drinking was calculated by combining the reports for the seven days of the week (sum of the 7 days).
  Minimum = 0; Maximum = none
  Sample score range: Minimum = 0; Maximum = 26
  Higher scores are worse outcomes
Time Frame: Baseline, 1 month follow-up, and 6-month follow up
Population: One participant was removed from the analyses due to unreliable reporting
Measure: Mean (Standard Deviation); unit: drinks per week
Arm/Group | eCHECKUP TO GO | Control
Number analyzed (Participants) | 173 | 137
drinks per week
  Basline | 4.14 (6.74) | 3.06 (6.39)
  1 Month Follow-Up: number analyzed (Participants) | 158 | 124
  1 Month Follow-Up | 2.92 (4.93) | 2.55 (5.32)
  6 Month Follow-Up: number analyzed (Participants) | 148 | 118
  6 Month Follow-Up | 2.23 (3.94) | 2.14 (5.04)

2. Primary Outcome: Peak Drinking Quantity
Description: Quantity ⁄Frequency ⁄Peak Questionnaire
  Peak drinking quantity was assessed with the question "What is the most number of drinks that you have consumed on any given night in the past month?"
  Minimum = 0; Maximum = none
  Sample score range: Minimum = 0; Maximum = 25
  Higher scores are worse outcomes
Time Frame: Baseline, 1 month follow-up, and 6-month follow up
Population: One participant was removed from the analyses due to unreliable reporting
Measure: Mean (Standard Deviation); unit: drinks
Arm/Group | eCHECKUP TO GO | Control
Number analyzed (Participants) | 173 | 137
drinks
  Baseline | 5.10 (6.01) | 2.81 (5.13)
  1 Month Follow-Up: number analyzed (Participants) | 158 | 124
  1 Month Follow-Up | 3.65 (4.48) | 2.53 (4.89)
  6 Month Follow-Up: number analyzed (Participants) | 148 | 118
  6 Month Follow-Up | 3.63 (4.86) | 2.40 (4.58)

3. Primary Outcome: Frequency of Alcohol Use
Description: Quantity ⁄Frequency ⁄Peak Questionnaire
  Frequency of alcohol use was assessed with the question "How often do you use alcohol?" with responses provided on an 8-point Likert scale with options ranging from "0" to "7" ("Do not drink alcohol" to "Every day"). Items were reverse scores so higher scores represent higher levels of drinking frequency.
  Minimum = 0; Maximum = 7
  Sample score range: Minimum = 0; Maximum = 7
  Higher scores are worse outcomes
Time Frame: Baseline, 1 month follow-up, and 6-month follow up
Population: One participant was removed from the analyses due to unreliable reporting
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | eCHECKUP TO GO | Control
Number analyzed (Participants) | 173 | 137
score on a scale
  Baseline | 3.71 (1.94) | 2.84 (1.91)
  1 Month Follow-Up: number analyzed (Participants) | 158 | 124
  1 Month Follow-Up | 3.61 (1.89) | 2.72 (1.81)
  6 Month Follow-Up: number analyzed (Participants) | 148 | 118
  6 Month Follow-Up | 3.41 (1.80) | 2.62 (1.77)

4. Primary Outcome: Blood Alcohol Concentration
Description: Blood alcohol concentration was calculated using the Widmark Formula (1932/1981); BAC = [Alcohol consumed in grams / (Body weight in grams x r)] x 100. In this formula, "r" is the gender constant.
  Minimum = 0; Maximum = none
  Sample score range: Minimum = 0; Maximum = .62
  Higher scores are worse outcomes
Time Frame: Baseline, 1 month follow-up, and 6-month follow up
Population: One participant was removed from the analyses due to unreliable reporting
Measure: Mean (Standard Deviation); unit: percentage of alcohol/100 ml of blood
Arm/Group | eCHECKUP TO GO | Control
Number analyzed (Participants) | 173 | 137
percentage of alcohol/100 ml of blood
  Baseline | .11 (.16) | .06 (.11)
  1 Month Follow-Up | .07 (.11) | .05 (.11)
  6 Month Follow-Up | .09 (.15) | .07 (.15)

5. Primary Outcome: Heavy Episodic Drinking
Description: Heavy Episodic Drinking is defined as having 5 or more drinks in a row for males and 3 or more for females in a 2 hour period in the past month. The number of drinks was based on research by Donovan (2009) establishing cut-points for children and adolescents.
  Participants were asked:
  "Males: Think back over the last two weeks. How many times have you had 5 or more drinks in a two hour period?" "Females: Think back over the last two weeks. How many times have you had 3 or more drinks in a two hour period?"
  Minimum = 0; Maximum = none
  Sample score range: Minimum = 0; Maximum = .76
  Higher scores are worse outcomes
Time Frame: Baseline, 1 month follow-up, and 6-month follow up
Population: One participant was removed from the analyses due to unreliable reporting
Measure: Mean (Standard Deviation); unit: binge drinking events
Arm/Group | eCHECKUP TO GO | Control
Number analyzed (Participants) | 173 | 137
binge drinking events
  Baseline | .89 (1.32) | .61 (1.32)
  1 Month Follow-Up: number analyzed (Participants) | 158 | 124
  1 Month Follow-Up | .73 (1.37) | .52 (1.14)
  6 Month Follow-Up: number analyzed (Participants) | 148 | 118
  6 Month Follow-Up | .66 (1.23) | .49 (1.22)

6. Secondary Outcome: Alcohol-Related Consequences
Description: Rutgers Alcohol Problems Inventory
  Alcohol-related consequences were measured using the Rutgers Alcohol Problems Inventory. The Rutgers Alcohol Problems Inventory is a 23-item scale. Participants were asked "How many times have the following scenarios happened to you while you were consuming alcohol or as a result of your drinking in the past 30 days." Responses were measured on a 5-point scale ranging from 0 (never) to 4 (more than 10 times). A total consequence score is created by summing the 23 items.
  Minimum = 0; Maximum = 92
  Sample score range: Minimum = 0; Maximum = 24
  Higher scores are worse outcomes
Time Frame: Baseline and 6-month follow up
Population: One participant was removed from the analyses due to unreliable reporting
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | eCHECKUP TO GO | Control
Number analyzed (Participants) | 173 | 137
score on a scale
  Baseline | 3.62 (5.52) | 2.35 (4.89)
  6 Month Follow-Up: number analyzed (Participants) | 148 | 118
  6 Month Follow-Up | 2.70 (4.97) | 1.45 (2.80)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | eCHECKUP TO GO | Control
All-Cause Mortality (participants affected / at risk) | 0/174 | 0/137
Serious Adverse Events (participants affected / at risk) | 0/174 | 0/137
Other Adverse Events (participants affected / at risk) | 0/174 | 0/137

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-01-27): https://cdn.clinicaltrials.gov/large-docs/18/NCT03613818/Prot_SAP_000.pdf